CLINICAL TRIAL: NCT00532727
Title: Triple Negative Trial: A Randomised Phase III Trial of Carboplatin Compared to Docetaxel for Patients With Metastatic or Recurrent Locally Advanced ER-, PR- and HER2- Breast Cancer.
Brief Title: Triple Negative Breast Cancer Trial
Acronym: TNT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: King's College London (Other); Cancer Research UK (Other); Breakthrough Breast Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2006/10003; ISRCTN97330959; Main REC: 07/Q0603/67; CTA: 22138/0004/001-0001; EudraCT Number: 2006-004470-26
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Triple Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Carboplatin
  Interventions: Drug: Carboplatin
- Arm B (Active Comparator): Docetaxel
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Carboplatin — AUC 6 every 3 weeks for six cycles (18 weeks)
  Arms: Arm A
Drug: Docetaxel — 100mg/m2 every 3 weeks for six cycles (18 weeks)
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine whether there is greater activity for carboplatin than a taxane standard of care (docetaxel) in women with ER-, PR- and HER2- breast cancer. The trial aims to recruit between 370 and 450 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ER-, PR-, primary breast cancer
* Histologically confirmed HER2- primary breast cancer
* Measurable confirmed metastatic or recurrent locally advanced disease unsuitable for local therapy but suitable for taxane chemotherapy
* Patients with stable, treated bain metastases will be eligible providing informed consent can be given and that other sites of measurable disease are present.
* Patients with bone metastases currently receiving bisphosphonates for palliation will be eligible providing informed consent can be given and that other sites of measurable disease are present
* ECOG Performance Status 0, 1, or 2
* Adequate haematology, biochemical indices (FBC, U & Es)
* LFTs = Normal bilirubin, AST and/or ALT = 3 x ULN if Alk Phos >5 x ULN (or an isolated elevation AST/ALT of ≤5 x ULN
* Adequate renal function - Creatinine clearance of >25mls per minute
* Written informed consent, able to comply with treatment and follow up

Exclusion Criteria:

* Original primary tumour or subsequent relapse known to be positive for any of ER, PR, or HER2 receptors
* Patients unfit for chemotherapy or those with neuropathy >grade 1 (sensory or motor)
* Known allergy to platinum compounds or to mannitol
* Known sensitivity to taxanes
* Patients with inoperable locally advanced disease suitable for local radiotherapy or an anthracycline containing regimen
* Previous chemotherapy for metastatic disease other than an anthracycline as in inclusion criteria above
* Previous exposure to a taxane in adjuvant chemotherapy within 12 months of trial entry
* Previous treatment with a taxane for recurrent locally advanced disease
* Previous treatment with a platinum chemotherapy drug
* LFTs = Abnormal bilirubin (> ULN), AST and/or ALT >3 X ULN and Alk Phos >5 x ULN (or an isolated elevation AST/ALT of >5 x ULN)
* Patients with a life expectancy of less than 3 months
* Previous malignancies other than adequately treated in situ carcinoma of the uterine cervix or basal or squamous call carcinoma of the skin, unless there has been a disease free interval of at least 10 years
* Previous or synchronous second breast cancer (unless also confirmed ER-, PR- and HER2-)
* Patients with bone limited disease
* Other serious uncontrolled medical conditions or concurrent medical illness likely to compromise life expectancy and/or the completion of trial therapy
* Pregnant, lactating or potentially childbearing women not using adequate contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Response: Response will be evaluated after three and six cycles of chemotherapy using modified Response Evaluation Criteria in Solid Tumours (RECIST) criteria, with appropriate clinical assessment and radiological investigations. | Time from start of treatment to 18 weeks

SECONDARY OUTCOMES:
Time to progression: this will be defined according to RECIST criteria and will be measured from the start of treatment until the confirmation of progression | Time from start of treatment until confirmation of progression
Progression free survival: this will be defined according to RECIST criteria and will be measured from the start of treatment until the confirmation of progression or death. | Time from start of treatment until confirmation of progression or death
Time to treatment failure: this will be defined as time from randomisation to discontinuation of protocol treatment for any reason, or progression of disease as defined by RECIST | Time from randomisation to discontinuation of protocol treatment for any reason, or progression of disease
Overall survival: this will be defined as time from randomisation until death from any cause in the intention to treat population | Time from randomisation until death from any cause
Toxicity will be assessed throughout the treatment period using the National Cancer Institute Common Terminology Criteria for Adverse Events version three (NCI CTCAE v3.0) | Time from start of treatment to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tutt, MB ChB, MRCP, FRCR, PhD, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Tutt A, Tovey H, Cheang MCU, Kernaghan S, Kilburn L, Gazinska P, Owen J, Abraham J, Barrett S, Barrett-Lee P, Brown R, Chan S, Dowsett M, Flanagan JM, Fox L, Grigoriadis A, Gutin A, Harper-Wynne C, Hatton MQ, Hoadley KA, Parikh J, Parker P, Perou CM, Roylance R, Shah V, Shaw A, Smith IE, Timms KM, Wardley AM, Wilson G, Gillett C, Lanchbury JS, Ashworth A, Rahman N, Harries M, Ellis P, Pinder SE, Bliss JM. Carboplatin in BRCA1/2-mutated and triple-negative breast cancer BRCAness subgroups: the TNT Trial. Nat Med. 2018 May;24(5):628-637. doi: 10.1038/s41591-018-0009-7. Epub 2018 Apr 30. PMID 29713086
- [Derived] Tovey H, Sipos O, Parker JS, Hoadley KA, Quist J, Kernaghan S, Kilburn L, Salgado R, Loi S, Kennedy RD, Roxanis I, Gazinska P, Pinder SE, Bliss J, Perou CM, Haider S, Grigoriadis A, Tutt A, Cheang MCU. Integrated Multimodal Analyses of DNA Damage Response and Immune Markers as Predictors of Response in Metastatic Triple-Negative Breast Cancer in the TNT Trial (NCT00532727). Clin Cancer Res. 2023 Sep 15;29(18):3691-3705. doi: 10.1158/1078-0432.CCR-23-0370. PMID 37574209
- [Derived] Sipos O, Tovey H, Quist J, Haider S, Nowinski S, Gazinska P, Kernaghan S, Toms C, Maguire S, Orr N, Linn SC, Owen J, Gillett C, Pinder SE, Bliss JM, Tutt A, Cheang MCU, Grigoriadis A. Assessment of structural chromosomal instability phenotypes as biomarkers of carboplatin response in triple negative breast cancer: the TNT trial. Ann Oncol. 2021 Jan;32(1):58-65. doi: 10.1016/j.annonc.2020.10.475. Epub 2020 Oct 21. PMID 33098992
- See also: Related Info — https://www.icr.ac.uk/our-research/centres-and-collaborations/centres-at-the-icr/clinical-trials-and-statistics-unit/clinical-trials/tnt